CLINICAL TRIAL: NCT03419078
Title: Route and Adequacy of Nutrition and Outcomes of Haematopoietic Cell Transplantation in Patients With Haematological Neoplasms
Brief Title: Nutrition and Outcomes of Hematopoietic Cell Transplantation (HCT)
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, JBeckerson, Haemato-Oncology Specialist Dietitian, Imperial College Healthcare NHS Trust
Other Study IDs: 15HH2638
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Allogeneic Stem Cell Transplant; Graft Versus Host Disease; Hematologic Malignancy; Stem Cell Transplant Complications
Keywords: enteral nutrition; parenteral nutrition; artificial nutrition support; non-relapse mortality; survival
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective case-note review to determine if nutrition via the enteral compared to the parenteral route results in better outcomes after haematopoietic cell transplantation.

DETAILED DESCRIPTION:
This is a retrospective case-note review of adults undergoing haematopoietic cell transplantation to treat a haematological malignancy who have been admitted to Hammersmith Hospital from 2000 to 2014. All patients receiving an allogeneic haematopoietic cell transplant from a matched sibling or identically matched unrelated donor will be included. We will record the route and assess the broad adequacy of nutritional intakes to determine if nutrition via the enteral compared to the parenteral route results in better outcomes after haematopoietic cell transplantation. Our outcomes are graft versus host disease incidence and severity, transplant related (early) mortality and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing their first HCT for a hematologic malignancy
* Undergoing HCT using a sibling or unrelated donor
* Undergoing HCT infusion between January 2000 and December 2014

Exclusion Criteria:

* HCT using umbilical cord blood donors
* HCT using haploidentical donors

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients aged 17 or above who underwent their first HCT for hematologic malignancy at Hammersmith Hospital, using a sibling or unrelated donor between January 2000 and December 2014
Sampling Method: Non-Probability Sample
Enrollment: 484 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Adequate Enteral Nutrition: Adequate nutrition in the period to engraftment after transplant, in those patients nourished orally or any patient that required 4 or more days of enteral tube feeding.
- Adequate Parenteral Nutrition: Patients that were adequately nourished during the period to engraftment after transplant, that received 4 or more days of parenteral nutrition.
- Inadequate Nutrition: Those with inadequate oral in take and a documented unmet need for artificial nutrition support for 4 or more days before engraftment.
Period: Overall Study
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Started | 245 | 148 | 91
Completed | 245 | 148 | 91
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition | Total
Number analyzed (Participants) | 245 | 148 | 91 | 484
Age, Customized [Count of Participants; unit: Participants]
  Age: <20 years | 3 | 5 | 2 | 10
  Age: 21-40 | 87 | 84 | 41 | 212
  Age: 41-60 | 134 | 53 | 40 | 227
  Age: >60 years | 21 | 6 | 8 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 47 | 36 | 179
  Male | 149 | 101 | 55 | 305
Diagnosis [Count of Participants; unit: Participants]
  Acute leukaemia | 73 | 57 | 28 | 158
  CML | 81 | 70 | 35 | 186
  Lymphoma & CLL MDS | 56 | 12 | 15 | 83
  MDS | 27 | 4 | 6 | 37
  Myeloma | 8 | 5 | 7 | 20
European Group for Blood and Marrow Transplantation (EBMT)disease risk [Count of Participants; unit: Participants] — The European Group for Blood and Marrow Transplantation (EBMT) risk score provides a simple tool to assess instantly chances and risks of hematopoietic SCT(HSCT) for an individual patient pre-transplant. Five factors, age of the patient, stage of the disease, time from diagnosis, donor type and donor recipient gender combination augment risk for an individual patient with increasing score from 0 as best to 7 as worst in an additive way. Early stage disease represents the better expected outcome.
  Participants
    Early staged | 110 | 75 | 44 | 229
    Intermediate staged | 70 | 47 | 22 | 139
    Late staged | 65 | 26 | 25 | 116
BMI (kg/m^2) [Count of Participants; unit: Participants]
  Underweight (less than 20) | 15 | 14 | 7 | 36
  Healthy (20 - 24.9) | 90 | 63 | 28 | 181
  Overweight (25 - 30) | 121 | 50 | 45 | 216
  Obese (over 30) | 19 | 21 | 11 | 51
Donor match [Count of Participants; unit: Participants]
  Matched sibling | 136 | 56 | 56 | 248
  Matched unrelated | 86 | 71 | 25 | 182
  Mismatch unrelated | 23 | 21 | 10 | 54
Conditioning [Count of Participants; unit: Participants]
  Myeloablative | 98 | 131 | 56 | 285
  Reduced intensity | 147 | 17 | 35 | 199
Previous autograft [Count of Participants; unit: Participants]
  yes | 26 | 9 | 12 | 47
  no | 219 | 139 | 79 | 437
Patient / Donor Sex [Count of Participants; unit: Participants]
  Other combination | 188 | 124 | 72 | 384
  Male / Female | 56 | 24 | 19 | 99
  Missing data | 1 | 0 | 0 | 1
Patient cytomegalovirus (CMV) serology [Count of Participants; unit: Participants]
  Positive | 100 | 71 | 31 | 202
  Negative | 142 | 77 | 58 | 277
  Missing data | 3 | 0 | 2 | 5
Donor CMV serology [Count of Participants; unit: Participants]
  Positive | 109 | 82 | 47 | 238
  Negative | 131 | 64 | 43 | 238
  Missing data | 5 | 2 | 1 | 8
Cells infused [Count of Participants; unit: Participants]
  PBSC | 184 | 88 | 54 | 326
  Bone marrow (BM) | 59 | 59 | 37 | 155
  PBSC + BM | 3 | 2 | 1 | 6
Cluster of differentiation 34 (CD34+) cells infused [Count of Participants; unit: Participants]
  Less than 4.00 x 10^6 | 40 | 46 | 29 | 115
  More than 3.99 x 10^6 | 173 | 87 | 53 | 313
  Missing data | 32 | 15 | 9 | 56
Era (years) [Count of Participants; unit: Participants]
  2000 - 2004 | 82 | 70 | 47 | 199
  2005 - 2009 | 78 | 42 | 18 | 138
  2010 - 2014 | 85 | 36 | 26 | 147
Hematopoietic cell transplant co-morbidity index (HCT-CI) [Count of Participants; unit: Participants] — The hematopoietic cell transplantation-comorbidity index (HCT-CI) is a comorbidity tool suited for recipients of HCT. The index has been shown to sensitively capture the prevalence and magnitude of severity of various organ impairments before HCT and to provide valuable prognostic information after HCT. The higher the comorbidities the worse the expected outcome.
  Participants
    0-1 | 130 | 70 | 50 | 250
    2-3 | 75 | 55 | 18 | 148
    more than 3 | 22 | 16 | 18 | 56
    missing data | 18 | 7 | 5 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Graft Versus Host Disease (GvHD) at Any Site (Grade II or Above) and Acute GvHD of the Gut of Any Grade
Description: Occurrence of acute GvHD at any site (grade II or above) and acute GvHD of the gut of any grade (graded according to standard criteria). Standard criteria to grade the severity of acute GvHD are quantification of rash, serum bilirubin and diarrhoea. These standard criteria have been developed and used for > 20 years by most transplant centres to improve comparability between publications.
Time Frame: 100 days after the date of hematopoietic cell infusion
Population: There were 439 and 438 evaluable cases respectively for acute GvHD grade II or greater and gastrointestinal acute GvHD of any grade after exclusion of patients that died before day 100 without acute GvHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Number analyzed (Participants) | 232 | 132 | 75
Participants
  Acute GvHD grade II-IV | 75 | 73 | 31
  Gut Acute GvHD any grade | 63 | 63 | 27

2. Primary Outcome: Non Relapse Mortality
Description: Defined as death without previous relapse
Time Frame: 100 days after the date of hematopoietic cell infusion
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Number analyzed (Participants) | 245 | 148 | 91
percentage of participants | 8.2 [5 to 12] | 17.6 [12 to 25] | 27.5 [20 to 38]

3. Secondary Outcome: Graft Versus Host Disease-free and Relapse-free Survival
Description: GvHD-free/relapse-free survival (GRFS). Events in GRFS included grade 3-4 acute GvHD, systemic therapy-requiring chronic GvHD, relapse, or death
Time Frame: 5 years after the date of hematopoietic cell infusion
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Number analyzed (Participants) | 245 | 148 | 91
percentage of participants | 39.183 [33 to 46] | 29.729 [22 to 39] | 27.472 [17 to 39]

4. Secondary Outcome: 5 Year Survival
Time Frame: 5 years after the date of hematopoietic cell infusion
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Number analyzed (Participants) | 245 | 148 | 91
percentage of participants | 53.877 [48 to 61] | 45.946 [38 to 55] | 41.758 [32 to 53]

ADVERSE EVENTS:
Arm/Group | Adequate Enteral Nutrition | Adequate Parenteral Nutrition | Inadequate Nutrition
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/148 | 0/91
Other Adverse Events (participants affected / at risk) | 0/245 | 0/148 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes